CLINICAL TRIAL: NCT00930839
Title: Exploring the Role of Prostaglandin D2 and the DP1 Receptor on Nicotinic Acid Induced Flushing
Brief Title: Role of Prostaglandins on Niacin-Induced Flushing
Status: Completed | Type: Observational
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Abbott (Industry)
Responsible Party: Aaron I. Vinik, MD, PhD, Eastern Virginia Medical School, Strelitz Diabetes Center
Other Study IDs: A10-597
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Flushing
Keywords: Niacin; Prostaglandin D2; Flushing; Nicotinic acid stimulated release of prostaglandin D2
MeSH Terms: conditions — Flushing | interventions — Niacin; Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin biopsies and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Controls: Normal, healthy controls, males and females, ages 30-80
  Interventions: Drug: Niacin and aspirin

INTERVENTIONS:
Drug: Niacin and aspirin — 1000 mg Niacin, 325 mg aspirin
  Other Names: Niaspan; Nicotinic acid

SUMMARY:
This study will focus on investigating the nicotinic acid stimulated release of prostaglandin D2 in normal controls. In subsequent studies, the investigators would like to further explore this pathway in people with type 2 diabetes. Enhanced blood flow (or flushing) may be compromised or exaggerated in type 2 diabetes particularly in those with impairment of autonomic function measured as the respiratory heart rate variability (HRV) of different frequencies reflecting the balance between the sympathetic and parasympathetic nervous systems. The investigators hypothesize that the vasodilatory effects induced by nicotinic acid will be different in glabrous and hairy skin and that autonomic imbalance may alter the response.

DETAILED DESCRIPTION:
The investigators propose that nicotinic acid (NA) stimulates release of prostaglandin D2 (PGD2). To fully understand this mechanism, the investigators will examine the systemic release of PGD2 and skin blood flow using laser Doppler (LDF) on the upper and lower limbs of healthy control subjects. The investigators will quantify and establish the effects of oral nicotinic acid (Niaspan®) given alone and in combination with aspirin on:

1. skin blood flow using laser Doppler (LDF) of glabrous and hairy skin of the forearm of healthy subjects
2. the severity and intensity of flushing using a visual analog scale, FAST tool, and whether aspirin is able to block the flushing response
3. the impact on sympathetic/parasympathetic balance using the various frequencies of heart rate variability (HRV) which reflect the contribution of the different divisions of the autonomic nervous system (ANS)
4. circulating levels of PGD2 and other neuropeptides to determine other mediators of the flushing response. This will allow us to conclude whether this pathway is intact and explore other non-DP1 vasodilatory mechanisms.
5. Langerhans cell density in epidermis and microvasculature using immunohistochemistry of Langerin (measured as CD1a) in 3 mm skin biopsies of volar and hairy surfaces of the forearm and hairy surface of the lateral aspect of proximal lower limb. To date, there is very little known about the density or distribution of Langerhans cells. The PGD2 receptor DP1 will be examined for its content in the epidermis using immunohistochemistry or RTPCR.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls ages 30-80

Exclusion Criteria:

1. Presence of type 1 diabetes or type 2 diabetes
2. Presence of clinically significant neuropathy, (Dyck stage >2b) defined by abnormal neurologic testing (neurologic physical exam, nerve conduction, autonomic and quantitative sensory tests)
3. History of major macrovascular events such as myocardial infarction or stroke within the past 3 months
4. Participation in another clinical trial concurrently or within 30 days prior to entry into this study.
5. Uncontrolled or untreated hypothyroidism as evidenced by TSH concentrations >4.8 uU/ml
6. Other serious medical conditions which, in the opinion of the investigator, would compromise the subject's participation in the study, including sensitivity to aspirin
7. Abnormalities of liver function defined as any liver enzymes (AST, ALT, SGPT, SGOT) greater than 3 times the upper limit of normal
8. History of NYHA Class IV congestive heart failure.
9. Allergy to Niaspan or aspirin
10. Use of drugs known to affect prostaglandin metabolism such as angiotensin converting enzyme inhibitors (ACE) inhibitors and angiotensin receptor blockers (ARBs) will be allowed with stable use for 3 months.
11. Pregnancy or breastfeeding
12. History of peptic ulcer disease
13. Current history of smoking

    -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal, healthy control subjects, males and females, ages 30-80
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy measures are skin perfusion measurements and neurological measures. | 30 minutes after administration of Niacin

SECONDARY OUTCOMES:
Secondary measures include blood chemistries | 15-30 min serial measurements

CONTACTS AND LOCATIONS:
Overall Officials: Aaron I Vinik, MD, PhD, Principal Investigator — Eastern Virginia Medical School, Strelitz Diabetes Center
Locations (1):
- Eastern Virgnia Medical School, Strelitz Diabetes Center, Norfolk, Virginia, United States